CLINICAL TRIAL: NCT03155724
Title: QP ExCELs: MultiPole Pacing (MPP) Sub-Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPP Sub-Study
Record Dates: First submitted 2017-05-15; First posted 2017-05-16 (Actual); Results first posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- MultiPole Pacing (Experimental): Traditional biventricular pacing CRT non-responders at the 3 or 6 month QP ExCELs study follow-up.
  Interventions: Device: MultiPole Pacing

INTERVENTIONS:
Device: MultiPole Pacing — CRT non-responders are programmed with MultiPole pacing ON.

SUMMARY:
The objective of this MultiPole Pacing (MPP) sub-study of the QP ExCELs study is to demonstrate that the MPP feature is effective by converting a percentage of cardiac resynchronization therapy (CRT) non-responders to responders. The MPP sub-study is a single-arm, multi-center, prospective trial within the ongoing QP ExCELs study (NCT02290028).

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in the ongoing QP ExCELs study
* Successfully implanted with a BIOTRONIK Ilivia 7 HF-T QP family CRT-D system, or future-marketed CRT-D system with the MPP feature. Successful implantation is defined as having at least two LV pacing vectors with a measured pacing threshold of ≤ 5.0 V @ any pulse width (allowing for a minimum 2.5 V safety margin) without phrenic nerve stimulation at the final programmed pacing output at the time of enrollment into the MPP sub-study.
* CRT Responder Assessment classification as "Worsened" or "Unchanged"
* Standard continuous biventricular (BiV) pacing from implant until the 6-Month QP ExCELs follow-up visit. (Implant to 3-Month QP ExCELs follow-up who qualify due to a Heart Failure (HF) hospitalization event)
* Able to understand the nature of the sub-study and give informed consent
* Available for an additional follow-up visit specific to the MPP sub-study at the investigational site
* No evidence of non-compliance to their ongoing commitment in the QP ExCELs study

Exclusion Criteria:

* Have a life expectancy of less than 6 months
* Expected to receive heart transplantation or ventricular assist device within 6 months
* Chronic atrial fibrillation
* Presence of another life-threatening, underlying illness separate from their cardiac disorder
* Received MPP pacing prior to enrolment into the MPP sub-study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (44):
- United States (44):
  - Thomas Hospital, Fairhope, Alabama
  - South Bay Electrophysiology, Inglewood, California
  - Eisenhower Desert Cardiology, Rancho Mirage, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Florida Hospital, Orlando, Florida
  - Orlando Health Heart Institute, Orlando, Florida
  - Florida Hospital Tampa Pepin Heart Institute, Tampa, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Parkview Physicians Group - Cardiology, Fort Wayne, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Hospital, Kansas City, Kansas
  - Baptist Health - Lexington, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Northeast Cardiology, Bangor, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Southcoast Health, Fall River, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - Cardiology Associates of North Mississippi, Tupelo, Mississippi
  - SSM Health St. Joseph Hospital - St. Charles, Saint Charles, Missouri
  - Mercy Clinic Cardiology, Springfield, Missouri
  - St. Louis Heart and Vascular, St Louis, Missouri
  - Glacier View Medical Research Institute, Cardiology, Kalispell, Montana
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - New York Presbyterian Queens, Flushing, New York
  - Weill Cornell Medicine, New York, New York
  - Mt. Sinai St. Luke's Hospital, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Westchester Medical Center, Valhalla, New York
  - Asheville Cardiology Associates, Asheville, North Carolina
  - Novant Health Winston-Salem Cardiology, Winston-Salem, North Carolina
  - Wake Forest Baptist Health Medical Center, Winston-Salem, North Carolina
  - Sanford Medical Center - Fargo, Fargo, North Dakota
  - University of Cincinnati, Cincinnati, Ohio
  - Temple Heart and Vascular Institute, Philadelphia, Pennsylvania
  - Upstate Cardiology, Greenville, South Carolina
  - UT Erlanger Cardiology, Chattanooga, Tennessee
  - Fort Worth Heart, Fort Worth, Texas
  - UT Health Science Center, The Woodlands, Texas
  - University of Utah Medical Center, Salt Lake City, Utah
  - UVM Medical, Burlington, Vermont

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MultiPole Pacing
Started | 53
Completed | 42
Not Completed | 11
Not completed — Death | 3
Not completed — Physician Decision | 1
Not completed — Study closure | 7

BASELINE CHARACTERISTICS:
Population: Baseline data collected from all participants enrolled, when available.
Arm/Group | MultiPole Pacing
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.3 (12.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 42
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height [Mean (Standard Deviation); unit: in] | 68.5 (4.0)
Weight [Mean (Standard Deviation); unit: Pounds] | 212.7 (52.69)

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Resynchronization Therapy (CRT) Responder Status With the MPP Feature
Description: Count of participants who are classified as "Improved", where responder classification is derived from a clinical composite score (CCS) based on changes in New York Heart Association (NYHA) class, Heart Failure (HF) hospitalization, and cardiovascular death.
  Responder classification at 6 months (evaluated compared to MPP Enrollment Visit) :
  * "Improved"
    * No HF hospitalization or cardiovascular death, AND
    * NYHA class is improved
  * "Unchanged"
    * No HF hospitalization or cardiovascular death, AND
    * NYHA class is unchanged
  * "Worsened"
    * HF hospitalization or cardiovascular death has occurred, OR
    * NYHA class is worsened
Time Frame: Enrollment to 6 Months
Population: Participants who have completed the MultiPole Pacing (MPP) Sub-study 6-Month follow-up visit or experienced a qualifying outcome event as of January 23, 2020.
Measure: Count of Participants; unit: Participants
Arm/Group | MultiPole Pacing
Number analyzed (Participants) | 45
Participants
  Improved | 16
  Unchanged | 23
  Worsened | 6
Statistical Analysis 1: Comparison: MultiPole Pacing; The primary endpoint 1 hypothesis was evaluated by performing an exact, binomial test comparing the binomial proportion of 'improved' patients to 3.0% with power of 80% and type 1 error (alpha) of 0.0224. A pre-planned interim analysis at 45 patients required a type 1 error (alpha) of 0.0026 to demonstrate significance; Test type: Superiority; p < 0.0001, Exact, binomial, one-sided

2. Secondary Outcome: Percentage of Participants Without MPP System Related Adverse Events Requiring Additional Invasive Intervention to Resolve at 6 Months.
Description: Evaluate adverse events that require additional invasive intervention to resolve specifically related to the MPP feature. These adverse events include any software issues related to MPP programming or any adverse event that occurs while MPP is enabled and that may be attributed to the use of the MPP feature. Outcome was evaluated as an adverse event free-rate (AEFR).
Time Frame: Enrollment to 6 Months
Population: Evaluable participants for Secondary Endpoint 1 include all participants who have been enrolled into the MPP Sub-Study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MultiPole Pacing
Number analyzed (Participants) | 53
percentage of participants | 100 [93.28 to 100.00]

3. Secondary Outcome: Clinical Composite Score (CCS) + Patient Global Assessment (PGA) Responder Status Utilizing a Modified CCS That Incorporates the PGA
Description: Evaluate a modified CCS, determining a responder classification based on changes in NYHA class, PGA, HF hospitalization, and cardiovascular death, where the PGA will ask participantss to assess how their overall status has changed since prior to receiving CRT therapy (markedly better, better, unchanged, worse, markedly worse).
  Modified responder classification (CCS + PGA) at 6 months (evaluated compared to MPP Enrollment Visit):
  * "Improved"
    * No HF hospitalization or cardiovascular death, AND
    * Neither NYHA class is worsened or PGA is worsened ("worse" or "markedly worse"), AND
    * NYHA class is improved or PGA is improved ("better" or "markedly better")
  * "Unchanged"
    * No HF hospitalization or cardiovascular death, AND
    * NYHA class is unchanged, AND
    * PGA is unchanged ("unchanged")
  * "Worsened"
    * HF hospitalization or cardiovascular death has occurred, OR
    * NYHA class is worsened or PGA is worsened ("worse" or "markedly worse")
Time Frame: Enrollment to 6 Months
Population: Participants who have completed the MPP Sub-Study 6-Month follow-up visit or experienced a qualifying outcome event as of January 23, 2020.
Measure: Count of Participants; unit: Participants
Arm/Group | MultiPole Pacing
Number analyzed (Participants) | 45
Participants
  Improved | 27
  Unchanged | 11
  Worsened | 7

4. Secondary Outcome: CCS Responder Status Utilizing an Expanded Responder Classification
Description: Evaluate a modified CCS with an expanded responder classification where "Improved" and "Unchanged" are considered responders.
  Responder classification at 6 months (evaluated compared to MPP Enrollment Visit) :
  * "Improved"
    * No HF hospitalization or cardiovascular death, AND
    * NYHA class is improved
  * "Unchanged"
    * No HF hospitalization or cardiovascular death, AND
    * NYHA class is unchanged
  * "Worsened"
    * HF hospitalization or cardiovascular death has occurred, OR
    * NYHA class is worsened
Time Frame: Enrollment to 6 Months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | MultiPole Pacing
Number analyzed (Participants) | 45
Participants
  Responder | 39
  Non-Responder | 6

ADVERSE EVENTS:
Time Frame: 6 months
Description: Sites were required to report any cardiovascular hospitalizations and any other hospitalizations in which cardiovascular symptoms occur on or before the date of the MPP 6-Month follow-up. These hospitalizations were categorized as Heart Failure Hospitalization, Non-Heart Failure Hospitalization, or if applicable, Non-system related/non-protocol defined. Extracardiac stimulation was assessed/categorized however other specific adverse event terms were not assessed.
Arm/Group | MultiPole Pacing
All-Cause Mortality (participants affected / at risk) | 3/53
Serious Adverse Events (participants affected / at risk) | 5/53
Other Adverse Events (participants affected / at risk) | 6/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MultiPole Pacing (N=53)
Heart Failure Hospitalization (Cardiac disorders) | 3
Non-Heart failure Hospitalization (General disorders) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MultiPole Pacing (N=53)
Non-system related/ Non Protocol-defined (Cardiac disorders) | 2 (2)
Extracardiac stimulation (Cardiac disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-06): https://cdn.clinicaltrials.gov/large-docs/24/NCT03155724/Prot_SAP_000.pdf